CLINICAL TRIAL: NCT00436514
Title: Colonoscopy by Videocapsuls Versus Standard Colonoscopy. Intra-individual Comparison for the Subject With a Medium or High Risk of Colorectal Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Pr Jean Paul Galmiche, CHU de Nantes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 06/12-L
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: patients; medium risk; asymptomatic; between 50 and 74 years old; high risk; case; history of neoplastic colic; cancers; polyps
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Polyps | interventions — Diet; Colonoscopy

INTERVENTIONS:
Behavioral: diet and absorption of ColoPEG — 4l of PEG during 2 days
Procedure: Colonoscopy with colic videocapsule — 2x 10mg Motilium, 2 Fleet Phospho soda (one is facultative) and 1 dulcolax (facultative)
Procedure: Standard colonoscopy — 1l of PEG the morning just before colonoscopy

SUMMARY:
Colorectal cancer is one of the most frequent and it prognosis is still serious. In France, diagnosis and screening applicated in numerous departements, and now in a path of generalization to the all country, is based on combination of searching blood into bowel movements (Haemoccult) for the screening of population with medium risk (age between 50 to 74 years old)and colonoscopy for the screening and diagnosis of pre-cancerous lesions for the patients with a high risk.Even if the efficiency of this strategy is proved, searching blood into the bowel movement by Haemoccult is still imperfect (a lot of false negative). Colonoscopy is not an ideal tool for screening. Indeed, its acceptability is not perfect and it constitute an invasive method, with complications, with a compulsory general anesthesia, implicating a high cost. The alternative of a screening method based on a non invasive method is required.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* patient able to give his informed consent
* No colorectal, intestinal inflammatory, ischemic or evolving infectious pathologies
* No signs of stenosis of small intestine or colon
* No contraindication to anesthesia
* No participation to an other clinical study
* Patient with and indication to colonoscopy for searching of a colorectal neoplasia during a screening program OR
* Patient for who a endoscopic following is required because of familial cases or personal cases of polyps or colorectal cancer

Exclusion Criteria:

* Presence of symptoms evocating an occlusive pathology
* Recent complicated colic diverticulosis
* No informed consent
* pregnancy or no use of efficient contraception treatment
* Patient with a pace-maker or others internal medical electronic device
* Evolved nephric or cardiac insufficiencies
* Hypersensibility to Fleet Phospho Soda (or one of the excipient), bisacodyl (or one of the excipient), motilium (or one of the excipient)
* Presence of a prolactinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Galmiche, MD, Study Director — Nantes University Hospital; Stanislas Chaussade, MD, Principal Investigator — Hôpital Cochin; Marie-Georges Lapalus, MD, Principal Investigator — Hospices Civils de Lyon; Christophe Cellier, MD, Principal Investigator — CHU Pompidou; Denis Heresbach, MD, Principal Investigator — Rennes University Hospital; Bernard Filoche, MD, Principal Investigator — CH de Saint Philibert; Vincent Maunoury, MD, Principal Investigator — CHU de Lille; Gerard Gay, MD, Principal Investigator — Central Hospital, Nancy, France; Thierry Barrioz, MD, Principal Investigator — Poitiers University Hospital; Emmanuel Ben Soussan, MD, Principal Investigator — University Hospital, Rouen; Dimitri Coumaros, MD, Principal Investigator — CHU de Strasbourg
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Sacher-Huvelin S, Coron E, Gaudric M, Planche L, Benamouzig R, Maunoury V, Filoche B, Frederic M, Saurin JC, Subtil C, Lecleire S, Cellier C, Coumaros D, Heresbach D, Galmiche JP. Colon capsule endoscopy vs. colonoscopy in patients at average or increased risk of colorectal cancer. Aliment Pharmacol Ther. 2010 Nov;32(9):1145-53. doi: 10.1111/j.1365-2036.2010.04458.x. Epub 2010 Sep 16. PMID 21039676